CLINICAL TRIAL: NCT04255147
Title: Helping Underdeveloped Lungs With Cells (HULC): Mesenchymal Stromal Cells in Extreme Preterm Infants at Risk of Developing Bronchopulmonary Dysplasia - Phase 1 Study
Brief Title: Cellular Therapy for Extreme Preterm Infants at Risk of Developing Bronchopulmonary Dysplasia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Ontario Institute of Regenerative Medicine (OIRM) (Unknown); Stem Cell Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HULC-1
Record Dates: First submitted 2020-01-14; First posted 2020-02-05 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Phase I clinical trial; Stem cells; Mesenchymal stromal cell; Bronchopulmonary Dysplasia; Preterm birth; Cell therapy
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mesenchymal Stromal Cell Therapy (Experimental): Patients are enrolled into one of three escalating dose panels based on the time of enrolment. The first three patients will receive 1 million cells/kg of body weight, the next three patients will receive 3 million cells/kg of body weight, and the final three patients will receive 10 million cells/kg of body weight. Progression through the escalating dose panels is subject to review by an independent Data Safety Monitoring Committee.
  Interventions: Biological: Allogeneic Umbilical Cord Tissue-Derived Mesenchymal Stromal Cells

INTERVENTIONS:
Biological: Allogeneic Umbilical Cord Tissue-Derived Mesenchymal Stromal Cells — Cryopreserved allogeneic umbilical cord tissue-derived mesenchymal stromal cells are thawed and administered intravenously.

SUMMARY:
Bronchopulmonary dysplasia (BPD) is a common and chronic lung disease that occurs in preterm infants following ventilator and oxygen therapy and is associated with long-term health consequences. Preclinical research shows that mesenchymal stromal cells (MSCs) can modify a number of pathophysiological processes that are central to the progression of BPD and thus present as a promising new treatment option. The main purpose of this Phase I study is to evaluate the safety of human umbilical cord tissue-derived MSCs in extremely preterm infants at risk of developing BPD.

DETAILED DESCRIPTION:
Complications of extreme preterm birth are the primary cause of mortality in children under the age of five. Bronchopulmonary dysplasia (BPD), the chronic lung disease that follows ventilator and oxygen therapy for acute respiratory failure, is the most common complication of extreme prematurity and contributes to life-long respiratory and neurological impairment. Currently, there is no effective treatment for BPD. The multi-factorial nature of BPD makes it challenging for traditional pharmacological therapies targeting a single pathway to have a major impact on outcome. Mesenchymal stromal cells (MSCs) may provide a promising new treatment avenue due to their pleiotropic effects that may prevent neonatal lung injury while promoting lung (and other organ) growth. A systematic review and meta-analysis of all preclinical studies testing MSCs in neonatal lung injury models provides strong evidence for the lung protective effect of MSCs. Additionally, studies in a large preclinical model of extreme prematurity and chronic lung injury suggest feasibility, safety and short-term hemodynamic benefit of intravenously delivered human umbilical cord tissue-derived MSCs (uc-MSC).

The aim of this study is to establish the safety, maximum feasible dose and feasibility of intravenously delivered allogeneic uc-MSCs in preterm infants at risk of developing BPD. This will be a Phase 1, open-label, single center, dose-escalating trial using a 3+3+3 design.

ELIGIBILITY:
A participant needs to meet all inclusion criteria between day of life 7-28 to be eligible:

Inclusion Criteria:

* Admission to The Ottawa Hospital (TOH) NICU - General Campus or Sunnybrook Health Sciences Centre NICU
* Gestational age at birth < 28 weeks
* Intubated on mechanical ventilation
* Fraction of inspired oxygen ≥ 30%
* Parents or substitute decision make must provide written informed consent

Exclusion Criteria:

* Severe congenital anomaly by antenatal ultrasound and physical examination
* Ongoing shock and severe sepsis (confirmed by positive blood or cerebrospinal fluid culture) as per attending physician
* Severe pulmonary hemorrhage
* Active pneumothorax (with chest tube in-situ)
* Hemodynamically significant PDA
* Participants with caregiver unable to speak English or French
* Patient i moribund, not expected to survive
* Planned to be extubated in the 24 hours after uc-MSC administration

Ages: 7 Days to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-11-06 (Actual); Study Completion 2033-11-06 (Estimated)

PRIMARY OUTCOMES:
Occurrence and rate of dose limiting toxicity | Up to 1 week following uc-MSC injection
  Dose limiting toxicity consists of the following events:
  * Death occurring within 24 hours of injection;
  * Pulmonary embolism defined as acute increase in right ventricular afterload (identified by serial targeted neonatal echocardiography) and signs of acute increased dead space ventilation (respiratory distress, increased PaCO2, increased minute ventilation) occurring within 24 hours of injection;
  * Hypersensitivity / anaphylactic to uc-MSCs defined as any severe systemic inflammatory response syndrome with negative blood culture not consistent with the overall clinical course of the infant occurring within 72 hours of injection;
  * Any other serious adverse event not expected in this patient population for which there is no alternative explanation but the administration of uc-MSCs, occurring within 1 week of injection.

SECONDARY OUTCOMES:
Rate of Death | From enrollment until discharge or 40 weeks corrected gestational age (whichever occurs first)
  Rate of death until discharge or 40 weeks corrected gestational age, whichever comes first
Occurrence of Other Severe Complications of Prematurity | From enrollment until discharge or 40 weeks corrected gestational age (whichever occurs first)
  * Blood culture-proven sepsis
  * Patent ductus arteriosus (treated medically or surgically)
  * Necrotizing enterocolitis
  * Isolated intestinal perforation
  * Retinopathy of prematurity requiring treatment
  * Severe intraventricular hemorrhage (≥ grade 3)
  * Cystic periventricular leukomalacia
FiO2 and Oxygen Index | From enrollment until discharge, 40 weeks corrected gestational age, or death (whichever occurs first)
  Measures of gas exchange
Need for Ventilatory Support | From enrollment until discharge, 40 weeks corrected gestational age, or death (whichever occurs first)
  * Time to extubation
  * Duration of mechanical ventilation
  * Duration of non-invasive positive pressure respiratory support
  * Duration of supplemental oxygen
Need for Postnatal Steroids | From enrollment until discharge, 40 weeks corrected gestational age, or death (whichever occurs first)
  This is a yes/no measure
Incidence and Severity of BPD | From enrollment until discharge, 40 weeks corrected gestational age, or death (whichever occurs first)
  Measured as mild, moderate, or severe
Rate of Survival Without (moderate or severe) BPD | From enrollment until 36 weeks corrected gestational age
  Measured according to the physiological definition of BPD (BPD at 36 weeks corrected age)
Changes in Pulmonary Hemodynamics | At enrollment, 48 hours following uc-MSC injection, 28 days of life, and 36 weeks corrected gestational age
  Targeted neonatal echocardiography to assess pulmonary hypertension using validated parameters
Biological Measure of Clinical Improvement | 72-96 hours following uc-MSC injection
  Markers of inflammation will be assessed in patient serum samples
Biological Measure of Lung Improvement | 72-96 hours following uc-MSC injection
  Biomarkers of lung improvement will be assessed in patient tracheal aspirate samples
Feasibility: Cell Administration | Day of life 7-28
  Successful recruitment and administration of cells to nine patients in 18 months
Feasibility: Recruitment Efficiency | Day of life 7-28
  * Proportion of potentially eligible patients that are successfully screened
  * Proportion of participants successfully screened who do not enroll (reason for failure to enroll will be recorded)
Feasibility: Recruitment Timing | Day of life 7-28
  * Median time from screening to enrollment
  * Median time from screening to cell administration
Feasibility: Participant Retainment | From enrollment until follow-up at 18-30 months-of-age
  * Proportion of patients that do not complete cell infusion
  * Proportion of patients enrolled that do not undergo scheduled follow-up
Bayley Scale of Infant and Toddler Development | 18-30 months-of-age
  Assessment of cognitive, language, and motor development
Long-term Safety Follow-Up | Ten years following follow-up visit
  Participant's overall health will be assessed through a questionnaire administered over the phone, once a year for 10 years
Animated Information Video | Day of life 7-28
  Characterize parental views of an animated MSC information video through brief semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Thébaud, MD, PhD, Principal Investigator — Ottawa Hospital Research Institute
Locations (2):
- Canada (2):
  - The Ottawa Hospital - General Campus, Gloucester, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size, the sharing of individual data has privacy and confidentiality implications.